CLINICAL TRIAL: NCT00585988
Title: Functional Recovery Following Hip Resurfacing or Total Hip Arthroplasty in Patients Matched By Age, Gender, and Activity Level
Brief Title: A Clinical Investigation of Recovery Following Hip Resurfacing or Total Hip Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 292-U-010
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Arthritis; Traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other)
  Interventions: Device: Hip Resurfacing System
- 2 (Other)
  Interventions: Device: M2a-Magnum™ Large Metal Articulation

INTERVENTIONS:
Device: Hip Resurfacing System — This arm will utilize a hip resurfacing system.
  Arms: 1
Device: M2a-Magnum™ Large Metal Articulation — This arm will utilize the M2a-Magnum™ implant system.
  Arms: 2

SUMMARY:
The primary purpose of this study is to compare early functional outcomes in patients undergoing hip resurfacing and total hip arthroplasty with the M2a-Magnum™ using more objective measures of function.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring hip arthroplasty

Exclusion Criteria:

* Patients with sensory, neurological, or general health conditions that alter perception of their limb in space
* Patients with vestibular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2009-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Functional Tests | 1 year